CLINICAL TRIAL: NCT02763189
Title: The Effects of Mentoring on Apnea Time While Using a Novel Fiber-optic Assisted Coaxial Endotracheal Tube Exchange Device
Brief Title: Effect of Mentoring on Endotracheal Tube Exchange Using a New Device
Acronym: FACETTE2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The device did not work well enough in its current form to continue the study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00037896
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2018-08

CONDITIONS: Effects of Training
Keywords: Mentoring; Endotracheal Tube Exchange; Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control group will study the learning material independently. 'Self-study'.
  Interventions: Other: Self-study
- Mentored (Experimental): Mentored group will study the learning materials and then receive expert mentoring
  Interventions: Other: Expert mentoring; Other: Self-study

INTERVENTIONS:
Other: Expert mentoring — Experts will provide personalized instructional review on how to use the new device for changing endotracheal tubes.
  Arms: Mentored
Other: Self-study — All subjects will receive self-study

SUMMARY:
The purpose of this pilot study is to compare the time it takes to change a breathing tube with a new device, performed by two different groups of anesthesiologists; one group will study on their own how to change the tube, while the second group will also receive expert training, before either group performs the procedure for the very first time. The Investigators predict the group who gets expert training will change the tube faster, and those investigators also need to learn how much faster, before moving to a larger study.

DETAILED DESCRIPTION:
After informed consent is obtained, two groups of randomized anesthesiologists will receive detailed instructional materials including a brochure to introduce the new device, a videotape showing how the device is used, a detailed slide show explaining each of the steps, and a checklist of the steps to perform during the exchange (E) in simulation. The Mentored group (M) will also receive expert instruction just before the procedure, while the Control group (C) will have the same amount of time to review the steps themselves. Next, they will perform the first exchange procedure (E1) while the pair of experts observe and measure the simulated patients' apnea time. The experts will then conduct a debriefing with the M group, while the C group will debrief themselves before both groups perform the exchange a second time (E2). Both groups will then receive debriefing by the experts. The apnea times and a performance assessment will be compared between M and C to determine the effects of expert training, and will also be compared within each group from E1 to E2, to determine the effect of experience on apnea time and performance. Finally, surveys conducted after E1 and E2, and before debriefing, will determine the participants' satisfaction with the new device. Data on apnea times will be used for a statistical power analysis to determine the size of a larger group necessary to show significant differences in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* physician airway management experts
* training in the skill of fiber-optic endoscopic intubation

Exclusion Criteria:

* non-physicians
* physicians without airway management expertise
* physicians without skill in fiber-optic endoscopic intubation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Olympio, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Apnea times will be shared at the conclusion of the study

REFERENCES:
- [Background] Hudes ET, Fisher JA, Guslitz B. Difficult endotracheal reintubations: a simple technique. Anesthesiology. 1986 Apr;64(4):515-7. doi: 10.1097/00000542-198604000-00020. No abstract available. PMID 3963460
- [Background] Olympio MA, Reinke B, Abramovich A.
- See also: APSF Newsletter Article by Dr. Olympio on Technology Training — http://www.apsf.org/newsletters/html/2006/fall/02training.htm
- See also: Product description of the novel tube exchanger used in this study. — http://www.wakeforestinnovations.com/technology-for-license/endotracheal-tube-exchanger/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Mentored
Started | 4 | 4
Completed | 4 | 2
Not Completed | 0 | 2
Not completed — Device failure | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Mentored | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Apnea Time
Description: Apnea time was measured in seconds from the time the ventilator was disconnected from the original endotracheal tube to the time the ventilator was connected to the new endotracheal tube immediately after procedure.
Time Frame: immediately after the procedure
Measure: Mean (Full Range); unit: seconds
Arm/Group | Control | Mentored
Number analyzed (Participants) | 4 | 4
seconds | 146 [129 to 164] | 111 [111 to 111]

2. Secondary Outcome: Performance Score
Description: The performance score is obtained form the performance Score Sheet that includes 15 actions, 1 point is given for each completed action. The minimum score is 0, the maximum score is 15. Higher scores relate to better performance.
Time Frame: immediately after the procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control | Mentored
Number analyzed (Participants) | 4 | 4
units on a scale | 11.75 [11 to 14] | 11 [9 to 14]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Control | Mentored
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Technical problems with the device used in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes